CLINICAL TRIAL: NCT04668781
Title: Improvement of Care of Patients Undergoing Pancreaticoduodenectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Principal Investigator, Piia Peltoniemi, M.D., Principal Investigator, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3169/2018
Record Dates: First submitted 2020-12-09; First posted 2020-12-16 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Diseases; Pancreas Cancer
Keywords: pancreaticoduodenectomy; fluid therapy; enhanced recovery after surgery (ERAS); postoperative complications
MeSH Terms: conditions — Pancreatic Diseases; Pancreatic Neoplasms; Postoperative Complications

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epidural analgesia (Active Comparator)
  Interventions: Procedure: Analgesia via epidural catheter
- Wound catheter analgesia (Experimental)
  Interventions: Procedure: Analgesia via wound catheter

INTERVENTIONS:
Procedure: Analgesia via epidural catheter — Ropivacain-infusion 2 mg/ml 1,25ml/h/10kg IBW (ideal body weight) is started to patients in the beginning of the surgery and is continued to POD 4. The rest of the treatment obey study protocol in both groups.
  Arms: Epidural analgesia
Procedure: Analgesia via wound catheter — Ropivacain 5 mg/ml 2,5ml/10kg IBW (ideal body weight) is given to patients in the end of the surgery. After that ropivacain-infusion 2mg/ml 1,25ml/h/10kg IBW is started to patients and is continued to POD 4. The rest of the treatment obey study protocol in both groups.
  Arms: Wound catheter analgesia

SUMMARY:
The study is a randomised controlled trial comparing the effectivity and impact of epidural analgesia and wound catheter analgesia in patients undergoing pancreaticoduodenectomy. The aim of the study is to examine whether there are a difference in perioperative fluid therapy and complication rates between the patients in epidural and wound catheter groups.

DETAILED DESCRIPTION:
All patients undergoing pancreaticoduodenectomy in Helsinki University Hospital are recruited in the study. Patients meeting the inclusion criteria and giving consent to participate the study will be randomised to whether epidural analgesia group or wound catheter analgesia group. Both groups receive additional analgesia with intravenous PCA-oxycodone (patient controlled analgesia).

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or over
* patients who undergo pancreaticoduodenectomy

Exclusion Criteria:

* patients to whom are made a major vascular reconstruction
* patients with significant comorbidities and inability to use PCA
* regural use of strong opioids or drugs preoperatively
* patients with severe chronic pain issues
* chronic atrial fibrillation
* patients who refuse to take part to the study

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-12-18 (Actual)

PRIMARY OUTCOMES:
The norepinephrine consumption | Postoperative day 0
  Norepinephrine consumption on POD 0

SECONDARY OUTCOMES:
Fluid volumes on PODs 0-4 | Postoperative days 0-4
  Intraoperative and postoperative fluid volumes
Oxycodone consumption | Postoperative days 1-4
  Intravenous PCA opioid consumption.
Hospital length of stay | Postoperative days 0-60
Postoperative complications | Postoperative days 0-90
  Clavien-Dindo complications (scale 0-5), pancreatic fistulas (ISGPF definition, grade A-C), postpancreatectomy hemorrage (IPGPS definition, grade A-C), delayed gastric emptying (ISGPS definition, grade A-C).
Reoperation rates | Postoperative days 0-90
Readmission rates | Postoperative days 0-90
Mortality | postoperative day 0-90

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Hospital, Helsinki, HUS, Finland

IPD SHARING:
Plan to Share IPD: No